CLINICAL TRIAL: NCT02537834
Title: An Open-Label, Multicenter Study to Evaluate 52-Week Long-Term Safety, Tolerability and Efficacy of Tofogliflozin With Glucagon-like Peptide-1(GLP-1) Analogue Treatment In Type 2 Diabetes Mellitus
Brief Title: Tofogliflozin GLP-1 Analogue Combination Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEBT02; TOFOGL07279 (Other: Sanofi)
Record Dates: First submitted 2015-08-25; First posted 2015-09-02 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-((4-ethylphenyl)methyl)-3',4',5',6'-tetrahydro-6'-(hydroxymethyl)spiro(isobenzofuran-1(3H),2'-(2H)pyran)-3',4',5'-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tofogliflozin ＋GLP-1 analogue (Experimental): Tofogliflozin administered once daily for 52 weeks. GLP-1 analogue administered as base treatment.
  Interventions: Drug: Tofogliflozin; Drug: GLP-1 analogue

INTERVENTIONS:
Drug: Tofogliflozin
  Other Names: DEBERZA; APLEWAY
Drug: GLP-1 analogue

SUMMARY:
An open-label, multicenter study to evaluate 52-week long-term safety, tolerability and efficacy of Tofogliflozin with GLP-1 analogue treatment in type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* The subject aged from 20 to 75 years old with type 2 diabetes mellitus(T2DM)
* The subject with hemoglobin A1c ≧7.5% - <10.5 %
* The subject who has been receiving a stable dose and regimen of GLP-1 analogue over 8 weeks before Screening test

Exclusion Criteria:

* The subject with type 1 diabetes mellitus
* The subject with Pregnancy or lactation
* The subject with Fasting Plasma Glucose ≧ 270 mg/dl
* The subject with history of metabolic acidosis, including diabetic ketoacidosis ,within 1 year prior to screening
* The subject with myocardial infarction, stroke, or heart failure requiring hospitalization or drug or alcohol abuse within the previous 6 months
* The subject with serum creatinine level greater than 2.0 mg/dL for men and 1.5 mg/dL for women
* The subject with aspartate aminotransferase(AST) or alanine aminotransferase(ALT) ≧ 2.5 times the upper limit of the reference range at the central laboratory test facility
* The subject has received treatment with another investigational product or non-approved drug 3 months before screening
* The subject with history of Tofogliflozin therapy
* The subject with estimated glomerular filtration rate of <30 mL/min/1.73 m^2
* The subject who frequently experiencing orthostatic hypotension
* The subject systolic blood pressure of ≧ 180 or mmHg of diastolic blood pressure of ≧ 100 mmHg
* The subject required a change in the dosing regiment for the following drugs within 4 weeks before screening : Lipid-lowering drug , Antihypertensive drug, Thyroid hormone drug , Uric acid lowering drug

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-08; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Assessed by Adverse Event and Adverse Drug Reaction | baseline and Week 52
Change from Baseline in HbA1c at 52 weeks | Week 52

SECONDARY OUTCOMES:
Change in Fasting plasma glucose | baseline and week 52
Change in Body Weight | baseline and week 52
Change in Blood pressure | baseline and week 52
Change in Uric Acid | baseline and week 52
Change in Total cholesterol | baseline and week 52
Change in HDL-C | baseline and week 52
Change in LDL-C | baseline and week 52
Change in non HDL-C | baseline and week 52
Change in Free Fatty Acid | baseline and week 52

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - Atsuta-ku, Aichi-ken
  - Minato-ku, Aichi-ken
  - Kisarazu, Chiba
  - Annaka, Gunma
  - Naka, Ibaraki
  - Sagamihara, Kanagawa
  - Kasaoka, Okayama-ken
  - Shimono, Tochigi
  - Adachi-ku, Tokyo
  - Chuo-ku, Tokyo
  - Mitaka, Tokyo

REFERENCES:
- [Result] Terauchi Y, Fujiwara H, Kurihara Y, Suganami H, Tamura M, Senda M, Gunji R, Kaku K. Long-term safety and efficacy of the sodium-glucose cotransporter 2 inhibitor, tofogliflozin, added on glucagon-like peptide-1 receptor agonist in Japanese patients with type 2 diabetes mellitus: A 52-week open-label, multicenter, post-marketing clinical study. J Diabetes Investig. 2019 Nov;10(6):1518-1526. doi: 10.1111/jdi.13066. Epub 2019 May 28. PMID 31033218
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31033218/